CLINICAL TRIAL: NCT06592911
Title: Multicentric Randomized Non-inferiority Study Examining the Effect of the Digital Medical Device Poppins Clinical for Cognitive and Musical Training in Addition to Bi-monthly Speech and Reading Therapy Sessions on the Reading and Writing Skills of Pediatric Participants With a Specific Learning Disability With Reading and/or Written Expression Deficit Compared With a Control Group Receiving Weekly Speech and Reading Therapy Sessions.
Brief Title: Examining the Effect of a Digital MD for Cognitive and Musical Training + Reduced Conventional SOC on the Reading and Writing Skills of Pediatric Participants With a Specific Learning Disability With Reading and/or Written Expression Deficit vs a Control Group Receiving Conventional SOC.
Acronym: POPPINS-02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poppins (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POPPINS-02
Record Dates: First submitted 2024-01-09; First posted 2024-09-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Learning Disorder, Specific; Learning Disability; Specific Learning Disorder, With Impairment in Reading; Dyslexia
MeSH Terms: conditions — Specific Learning Disorder; Learning Disabilities; Dyslexia

STUDY DESIGN:
Intervention Model Description: Multicentric randomized non-inferiority study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (No Intervention): 1 session of speech and reading therapy weekly, no use of the medical device Poppins Clinical
- EXPERIMENTAL (Experimental): Reduced speech and reading therapy sessions (1 session every 2 weeks) and use of the medical device Poppins Clinical
  Interventions: Device: Poppins Clinical

INTERVENTIONS:
Device: Poppins Clinical — Poppins Clinical is a software as a medical device that combines a musical and cognitive training program and written language training program.
  Arms: EXPERIMENTAL

SUMMARY:
Poppins-02 is a multicentric randomized non-inferiority study examining the effect of the digital medical device Poppins Clinical for cognitive and musical training in addition to bi-monthly speech and reading therapy sessions on the reading and writing skills of pediatric participants with a specific learning disability with reading and/or written expression deficit.

Participants will be assigned randomly either to an experimental group that will use the medical device in combination with reduced speech and reading therapy sessions (1 session each 2 weeks) or to the control group receiving conventional standard of care, i.e. 1 speech and reading therapy sessions per week.

DETAILED DESCRIPTION:
The study is a multicentric randomized non-inferiority clinical trial that has the aim to evaluate the impact of the digital medical device Poppins Clinical in addition to reduced speech and reading therapy sessions on children aged 7 to 11 years on their reading and writing skills.

Poppins Clinical is a software as a medical device (saMD) that combines a musical and cognitive training program and a written language training program. It is intended to provide a therapeutic rehabilitation for children with Specific Learning Disorders (SLD) with reading deficit. Poppins Clinical saMD operates on a tablet or smartphone and is designed to offer a fun and interactive gaming experience for children in form of a serious game.

The POPPINS-02 study thus proposes to include two patient arms:

* The experimental arm benefiting from Poppins Clinical training during 12 weeks in addition to reduced conventional speech and reading therapy (1 session each 2 weeks),
* The control arm having only conventional speech and reading therapy (1 session per week) during 12 weeks.

A randomization list will be generated, directing patients to the experimental or control arm, and informing parents, the patient, and the speech and reading therapist after the first pre-test. The investigator and his team will be blinded to the patient allocation group. It is therefore a single-blind study since parents, patients, and speech and reading therapists will be aware of the randomization.

In the experimental group, patients will have access to training with Poppins Clinical for 5 sessions per week, each session lasting approximately 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLD with reading deficit, based on a speech-language assessment. SLD with reading deficit is defined in the Diagnostic and Statistical Manual of Mental Disorders (DSM-5-TR, 2022). The speech-language assessment should consist of at least three reading and/or transcription tests with a SD (standard deviation) of at least - 1.4 or a result below the 20th percentile or two reading and/or transcription tests with a SD of at least - 2 SD or a results below the 10th percentile;
* Subject aged between 7 and 11, enrolled from CE1 to CM2;
* Subject receiving speech and reading therapy for less than 2 years, receiving speech and reading therapy for written language for less than 2 years, with a maximum treatment frequency of one session per week, either for at least 3 months for children followed for more than 3 months, or for the duration of the treatment for children followed for less than 3 months.;
* French mother tongue or French bilingualism at home and more than 3 years schooling in France;
* Tablet or smartphone available at home;
* Subject affiliated to the French National Insurance (Sécurité Sociale);
* Subject and parental/legal guardians consent to participate, and commitment to follow the protocol.

Exclusion Criteria:

* Subject has previously used Poppins Clinical or a previous version (Mila-Learn);
* Unstabilized chronic illness (at investigator's discretion);
* Participants with autism spectrum disorders or documented intellectual disabilities;
* Vision or Hearing difficulties preventing the use of the tablet or smartphone;
* Any condition that, in the opinion of the investigator, may prevent the patient from participating in the trial
* Participant actively participating in an interventional study that may affect results.
* Concurrent participation of any other family member in the same clinical trial

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 306 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-01-29 (Actual); Study Completion 2026-01-29 (Actual)

PRIMARY OUTCOMES:
Evaluate the non-inferiority of Poppins Clinical as a complement to reduced speech and reading therapy compared to only speech and reading therapy. | 12 weeks
  This endpoint evaluates the non-inferiority on reading abilities using a word reading task measured by the EVALEO 2-minute word reading test (EVAL2M) and measuring the number of correctly read words.

SECONDARY OUTCOMES:
Secondary safety objective | 12 weeks
  any adverse events will be collected from participants.
  Evaluation of adverse events reported by participants
Secondary objective 1: Evaluate the effect of adding Poppins Clinical on reading abilities in terms of speed (non-inferiority) | 12 weeks
  This endpoint evaluates the non-inferiority on reading abilities using a word reading task measured by the EVALEO 2-minute word reading test (EVAL2M) and measuring the number of read words.
Secondary objective 2: Evaluate the effect of adding Poppins Clinical on text reading skills (non-inferiority) | 12 weeks
  This endpoint evaluates the effect of the addition of Poppins Clinical on word reading skills in terms of speed and accuracy as assessed by a text reading test (Alouette).
Secondary objective 3: description and evaluation of the coast associated to children's treatment | 12 weeks
  This endpoint evaluates the coasts related to the medical care between the two groups, based on the number of treatment sessions, cost per session, cost of the medical device and travel cost, using a custom-made questionnaire
Secondary objective 4: Evaluation of the effect of adding Poppins Clinical on the parents' stress level between the two groups (EXPE/CONT) (non-inferiority) | 12 weeks
  This endpoint examines the impact of adding Poppins Clinical on parents' stress levels, measured using the parenting stress index short form
Secondary objective 5: Description and comparison of the effect of adding Poppins Clinical on the parents' quality of life between the two groups (EXPE/CONT) (non-inferiority) | 12 weeks
  This endpoint examines the impact of adding Poppins Clinical on parents' quality of life, measured using the EQ-5D-5L quality of life questionnaire
Secondary outcome 6: evaluate the effect of adding Poppins Clinical on meta-phonological skills between the two groups (EXPE/CONT) (non-inferiority) | 12 weeks
  This endpoint evaluates the effect of adding Poppins Clinical on meta-phonological skills as assessed by the BALE phoneme suppression test (correct answers score)
Secondary objective 7: Evaluate the effect of adding Poppins Clinical on text comprehension (non-inferiority) | 12 weeks
  This endpoint evaluates at the effect of adding Poppins Clinical on text comprehension assessed using the computerized adaptable test battery (BMT-i)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Pitié-Salpêtrière, Paris, Paris 75013, Paris
  - Hôpital Henri Laborit Poitiers, 86000, Poitiers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grossard C, Descamps M, Cadoni S, Pellerin H, Vonthron F, Xavier J, Falissard B, Cohen D. Assessing the Noninferiority of a Rhythm and Language Training Serious Game Combined With Speech Therapy Versus Speech Therapy Care for Children With Dyslexia: Protocol for an Investigator-Blinded Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 3;14:e71326. doi: 10.2196/71326. PMID 40179385